CLINICAL TRIAL: NCT05872438
Title: Evaluation of Multisite Sampling to Detect C. Trachomatis or N. Gonorrheae Compared With Vaginal Sampling in Women at Risk for Sexually Transmitted Infections (STI)
Brief Title: Evaluation of Multisite Sampling to Detect C. Trachomatis or N. Gonorrheae Compared With Vaginal Sampling in Women at Risk for Sexually Transmitted Infections
Acronym: SIST'RS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2022-16
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Sexually Transmitted Infection
Keywords: Sexually Transmitted Infection; PCR; C. trachomatis; N. gonorrhoeae; Screening
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Comparison of screening for two hypothesis:
  How many and what percentage of additional STI are diagnosed with the 3 sites sampling compared to the vaginal sampling alone?
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multisite sampling (Other): Vaginal, Oral and anal sampling for all participants
  Interventions: Diagnostic Test: Vaginal, Oral and anal sampling

INTERVENTIONS:
Diagnostic Test: Vaginal, Oral and anal sampling — The patients will take the samples themselves from the 3 sites (vaginal, anal and oral self-sampling) using standard swabs (brand). The sample will immediately be placed in the transport medium in each of the 3 Sigma VCM tubes labeled by the patient, depending on the collection site. The study nurse will register the inclusion of patients, identify the tubes, collect information and send them to the local laboratory for the PCR to be performed.

SUMMARY:
Screening for STIs in MSM is based on multisite samples: urine, anal and oral for PCR targeting C. trachomatis, N. gonorrhoeae, M. genitalium and T. vaginalis, whereas only vaginal self-sampling is recommended in women.

Recent publications and observations suggest that a substantial number of STIs are under diagnosed with the current recommendations.

The main objective of the study is to assess the number and percentage of additional C. trachomatis and N. gonorrhoeae infections diagnosed by a multiple sampling strategy in women, particularly when the vaginal sampling is negative The secondary objective will assess the acceptability of anal and oropharyngeal self-sampling relative to vaginal self-sampling in women.

DETAILED DESCRIPTION:
1500 women will be included in 5 different screening STIs centers in France based of the prevalence of STIs in this population (10% C. trachomatis) and the hypothesis that this new strategy allows to detect 20% more underdiagnosed STIs The sequential recruitment will concern women attending at one of the 5 STIs screening centers, whether they are symptomatic or not. If they agree to participate in the study, the patients will take the samples themselves from the 3 sites (vaginal, anal and oral self-sampling) using standard swabs (brand). The sample will immediately be placed in the transport medium in each of the 3 Sigma VCM tubes labeled by the patient, depending on the collection site. The study nurse will register the inclusion of patients, identify the tubes, collect information and send them to the local laboratory for the PCR to be performed. The study will be continued until the number of patients to be included for each of the centers is obtained. The anonymized data will be entered on an Excel database. The results of the PCRs will be collected a posteriori by the IDEs to populate the database. The PCR result will be given both qualitatively (positive/negative) and CT value for C. trachomatis and N. gonorrhoeae infections.

ELIGIBILITY:
Inclusion Criteria:

* Women coming for STI screening at a Cegidd
* Asymptomatic or not
* Women aged at least 18 years
* Having given her consent to participate

Exclusion Criteria:

* Patient having received antibiotic treatment covering C.trachomatis and N.gonorrheae in the month preceding the screening
* Patient under guardianship or curatorship
* Patient under legal protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Detectability of STIs in women on multisite samples | Baseline
  Number and percentage percentage of additional STI diagnosed with the 3 sites sampling compared to the vaginal sampling alone

SECONDARY OUTCOMES:
Percentage of women accepting anal and oropharyngeal self-sampling | Baseline
  acceptability of anal and oropharyngeal self-sampling relative to vaginal self-sampling in women

CONTACTS AND LOCATIONS:
Overall Officials: Julienne EFFA, Dr, Principal Investigator — CHU d'Orléans
Locations (7):
- France (7):
  - CeGIDD, Orléans
  - CHRU de POITIERS, Poitiers
  - Centre Hospitalier de Cornouaille, Quimper
  - CH de Saint Nazaire, Saint-Nazaire
  - CHU de STRASBOURG, Strasbourg
  - CHU de Tours, Tours
  - Centre Hospitalier de Vierzon, Vierzon

REFERENCES:
- [Background] Prazuck T, Lanotte P, Le Moal G, Hocqueloux L, Sunder S, Catroux M, Garcia M, Perfezou P, Gras G, Plouzeau C, Leveque N, Beby-Defaux A. Pooling Rectal, Pharyngeal, and Urine Samples to Detect Neisseria gonorrhoeae, Chlamydia trachomatis, and Mycoplasma genitalium Using Multiplex Polymerase Chain Reaction Is as Effective as Single-Site Testing for Men Who Have Sex With Men. Open Forum Infect Dis. 2022 Oct 31;9(10):ofac496. doi: 10.1093/ofid/ofac496. eCollection 2022 Oct. PMID 36324326
- [Background] Verougstraete N, Verbeke V, De Canniere AS, Simons C, Padalko E, Coorevits L. To pool or not to pool? Screening of Chlamydia trachomatis and Neisseria gonorrhoeae in female sex workers: pooled versus single-site testing. Sex Transm Infect. 2020 Sep;96(6):417-421. doi: 10.1136/sextrans-2019-054357. Epub 2020 May 13. PMID 32404400
- [Background] Lunny C, Taylor D, Hoang L, Wong T, Gilbert M, Lester R, Krajden M, Ogilvie G. Self-Collected versus Clinician-Collected Sampling for Chlamydia and Gonorrhea Screening: A Systemic Review and Meta-Analysis. PLoS One. 2015 Jul 13;10(7):e0132776. doi: 10.1371/journal.pone.0132776. eCollection 2015. PMID 26168051
- [Background] Alexander S, Ison C, Parry J, Llewellyn C, Wayal S, Richardson D, Phillips A, Smith H, Fisher M; Brighton Home Sampling Kits Steering Group. Self-taken pharyngeal and rectal swabs are appropriate for the detection of Chlamydia trachomatis and Neisseria gonorrhoeae in asymptomatic men who have sex with men. Sex Transm Infect. 2008 Nov;84(6):488-92. doi: 10.1136/sti.2008.031443. PMID 19028953
- [Background] Wayal S, Llewellyn C, Smith H, Hankins M, Phillips A, Richardson D, Fisher M; Home Sampling Kit Project Steering Group. Self-sampling for oropharyngeal and rectal specimens to screen for sexually transmitted infections: acceptability among men who have sex with men. Sex Transm Infect. 2009 Feb;85(1):60-4. doi: 10.1136/sti.2008.032193. Epub 2008 Aug 15. PMID 18708480
- See also: World Health Organization. Sexually transmitted infections — https://www.who.int/news-room/fact-sheets/detail/sexually-transmitted-infections-(stis)